CLINICAL TRIAL: NCT00243269
Title: Acupressure and Relaxation for Nausea Control
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Joseph Roscoe, Research Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: U2905
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2010-03

CONDITIONS: Nausea
Keywords: nausea, acupressure bands, relaxation
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Sham Comparator): Expectancy neutral handout and expectancy neutral tape
  Interventions: Behavioral: Acupressure expectancy enhancement
- 2 (Experimental): Expectancy enhancing handout and expectancy neutral tape
  Interventions: Behavioral: Acupressure expectancy enhancement
- 3 (Experimental): Expectancy neutral handout and expectancy enhancing tape
  Interventions: Behavioral: Acupressure expectancy enhancement
- 4 (Experimental): Expectancy enhancing handout and expectancy enhancing tape
  Interventions: Behavioral: Acupressure expectancy enhancement

INTERVENTIONS:
Behavioral: Acupressure expectancy enhancement — This study hypothesizes that patients receiving efficacy enhancing information about the acupressure bands will expect less treatment-related nausea, which will subsequently result in less treatment-related nausea compared to patients who do not receive such information.
  This study extends prior research by utilizing a randomized controlled trial in a clinical environment to examine the efficacy of an intervention that is specifically designed to reduce patients' response expectancies concerning nausea development from cancer treatments, and, thereby, reduce nausea.
  Other Names: 1 - Control handout and control tape; 2 - Active handout and control tape; 3 - Control handout and active tape; 4 - Active handout and active tape

SUMMARY:
This study hypothesizes that patients receiving efficacy enhancing information about the acupressure bands will expect less treatment-related nausea, which will subsequently result in less treatment-related nausea compared to patients who do not receive such information.

This study extends prior research by utilizing a randomized controlled trial in a clinical environment to examine the efficacy of an intervention that is specifically designed to reduce patients' response expectancies concerning nausea development from cancer treatments, and, thereby, reduce nausea.

The objectives of this study are as follow:

1. To provide preliminary data on whether a two-tiered strategy to increase patients' expectancies for nausea prevention and/or management will result in reduced chemotherapy-induced nausea.
2. To provide preliminary data on whether a two-tiered strategy to increase patients' expectancies for nausea prevention and/or management will result in increased health-related quality of life (HRQL) in patients receiving emetogenic chemotherapy.

To provide preliminary data on whether a two-tiered strategy to increase patients' expectancies for nausea prevention and/or management is more effective than a single-tiered strategy in reducing chemotherapy- induced nausea.

DETAILED DESCRIPTION:
This study hypothesizes that patients receiving efficacy enhancing information about the acupressure bands will expect less treatment-related nausea, which will subsequently result in less treatment-related nausea compared to patients who do not receive such information.

This study extends prior research by utilizing a randomized controlled trial in a clinical environment to examine the efficacy of an intervention that is specifically designed to reduce patients' response expectancies concerning nausea development from cancer treatments, and, thereby, reduce nausea.

The objectives of this study are as follow:

1. To provide preliminary data on whether a two-tiered strategy to increase patients' expectancies for nausea prevention and/or management will result in reduced chemotherapy-induced nausea.
2. To provide preliminary data on whether a two-tiered strategy to increase patients' expectancies for nausea prevention and/or management will result in increased health-related quality of life (HRQL) in patients receiving emetogenic chemotherapy.

To provide preliminary data on whether a two-tiered strategy to increase patients' expectancies for nausea prevention and/or management is more effective than a single-tiered strategy in reducing chemotherapy- induced nausea.

The study contains the following arms:

1. Control handout and control tape.
2. Active handout and control tape.
3. Control handout and active tape.
4. Active handout and active tape.

ELIGIBILITY:
Inclusion Criteria:

1) Have a diagnosis of breast cancer. 2) Be scheduled to receive a chemotherapy treatment containing doxorubicin (any dose) without concurrent radiotherapy or interferon. (Note: Chemotherapy agents in addition to doxorubicin may be given.) 3) Be 18 years of age or older. 3) Be chemotherapy naïve. 5) Be a female.

Exclusion Criteria:

1) Have clinical evidence of lymphedema, current bowel obstruction, or symptomatic brain metastases, as determined by their treating oncologist.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-11; Primary Completion 2009-05 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Roscoe, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester James P. Wilmot Cancer Center, Rochester, New York, United States

REFERENCES:
- [Result] Roscoe JA, O'Neill M, Jean-Pierre P, Heckler CE, Kaptchuk TJ, Bushunow P, Shayne M, Huston A, Qazi R, Smith B. An exploratory study on the effects of an expectancy manipulation on chemotherapy-related nausea. J Pain Symptom Manage. 2010 Sep;40(3):379-90. doi: 10.1016/j.jpainsymman.2009.12.024. Epub 2010 Jun 25. PMID 20579837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at three cancer clinics from Feb. 6, 2006 to April 23, 2009
Groups:
- Control Handout and Control Tape.: Patients received two acupressure bands. Patients received an expectancy-neutral handout that simply thanked them for participating in the study. The wording of the letter was, "Thank you for agreeing to participate in this study regarding the use of acupressure bands to control chemotherapy-related nausea. The information you will provide is extremely valuable. It is only with the assistance of individuals, like you, who are willing to give their time that we can learn new ways to better control the side effects of cancer treatment. Wear the acupressure bands for up to five days, if helpful, to prevent or alleviate nausea. We are very appreciative of your contribution to this study." Patients received an expectancy-neutral relaxation CD that was about 12 minutes in length and utilized guided imagery in which the individual visualized pleasant, soothing images or scenes while relaxed.
- Active Handout and Control Tape.: Patients received two acupressure bands.
  Patients received an expectancy-enhancing handout to enhance expected acupressure band efficacy. It was printed on Cancer Center letterhead and signed by a medical oncologist and two of the study investigators. The handout presented a very positive (and truthful) interpretation of the data from two prior acupressure band studies. Patients also received a medical prescription instructing them to use the acupressure bands for relief of nausea. The prescription was signed by a medical oncologist and had the instruction, "Wear Seabands for up to five days as needed to prevent or alleviate nausea." Patients' names were not on the prescription.
  Patients received an expectancy-neutral relaxation CD that was about 12 minutes in length and utilized guided imagery in which the individual visualized pleasant, soothing images or scenes while relaxed.
- Control Handout and Active Tape.: Patients received two acupressure bands. Patients received the same expectancy-neutral handout given to patients in Arm 1.
  Patients received the same relaxation CD as patients in the control condition with additional language inserted concerning efficacy of the acupressure bands and control of nausea. This additional language is under one minute in length and intended to strengthen patients' beliefs that the acupressure bands would be effective by focusing patients' attention on how effective the acupressure bands have been in reducing or eliminating nausea for other patients. In addition, it was suggested that since the acupressure bands were helpful to others, they might be helpful to them as well.
- Active Handout and Active Tape.: Patients received two acupressure bands. Patients received the same expectancy- enhancing handout given to patients in Arm 1.
  Patients received the same expectancy-enhancing CD given to patients in Arm 3.
Period: Overall Study
Arm/Group | Control Handout and Control Tape. | Active Handout and Control Tape. | Control Handout and Active Tape. | Active Handout and Active Tape.
Started | 31 | 11 | 12 | 29
Completed | 28 | 10 | 11 | 25
Not Completed | 3 | 1 | 1 | 4
Not completed — Protocol Violation | 2 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Handout and Control Tape. | Active Handout and Control Tape. | Control Handout and Active Tape. | Active Handout and Active Tape. | Total
Number analyzed (Participants) | 31 | 11 | 12 | 29 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 9 | 11 | 24 | 73
  >=65 years | 2 | 2 | 1 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (10.5) | 53.9 (9.4) | 49.1 (11.1) | 55.4 (9.9) | 51.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 11 | 12 | 29 | 83
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 11 | 12 | 29 | 83

OUTCOME MEASURES:

1. Primary Outcome: Five-day Nausea Diary
Description: Nausea was measured using a five-day patient report diary. Each day was divided into 4 sections: morning, afternoon, evening, and night. Patients reported severity of nausea for each period daily. Severity of nausea was assessed on a 7-point rating scale, anchored at one end by 1 = "Not at all nauseated" and at the other end by 7 = "Extremely nauseated." The description "Moderately nauseated" was centered on the scale below the 4. Average Nausea was the mean severity for the 20 reporting periods.
Time Frame: Five days
Population: All patients who did not have protocol violations who provided evaluable data were included in the analyses. No data imputation was used.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Control Handout and Control Tape. | Active Handout and Control Tape. | Control Handout and Active Tape. | Active Handout and Active Tape.
Number analyzed (Participants) | 28 | 10 | 11 | 25
Units on scale | 2.0 (1.1) | 2.1 (1.7) | 2.1 (0.9) | 1.9 (1.1)
Statistical Analysis 1: Comparison: Control Handout and Control Tape. vs Active Handout and Control Tape. vs Control Handout and Active Tape. vs Active Handout and Active Tape; The primary analyses consisted of calculating means and standard deviations on nausea for the four study arms to generate an effect size estimate for a later R01. We also planned to use a 2 x 2 (i.e., two levels of expectancy CDs and two levels of expectancy handouts) full factorial analysis of variance (ANOVA) to examine the efficacy of these two methods of expectancy enhancement in reducing Average Nausea as well as any interaction effects; Test type: Superiority or Other; p = 0.932, ANOVA

2. Secondary Outcome: Health Related Quality of Life
Description: Health-Related Quality of Life was assessed using the Functional Assessment of Cancer Therapy Scale - General (FACT-G). The FACT-G is a 28-item scale developed specifically for use in cancer clinical trials. Possible scores range from a low of 0 to a high of 112. Along with a total score representing HRQL, there are psychometrically validated subscales of physical, functional, social, and cognitive-emotional status. It has become one of the most commonly used measures in oncology, and we have used this scale in our previous studies.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Control Handout and Control Tape. | Active Handout and Control Tape. | Control Handout and Active Tape. | Active Handout and Active Tape.
Number analyzed (Participants) | 28 | 10 | 11 | 25
Units on scale | 75.2 (15.2) | 74.6 (14.9) | 70.9 (13.6) | 75.9 (17.2)
Statistical Analysis 1: Comparison: Control Handout and Control Tape. vs Active Handout and Control Tape. vs Control Handout and Active Tape. vs Active Handout and Active Tape; ANOVA to compare means of the four groups was used; Test type: Superiority or Other; p = 0.84, ANOVA

ADVERSE EVENTS:
Arm/Group | Control Handout and Control Tape. | Active Handout and Control Tape. | Control Handout and Active Tape. | Active Handout and Active Tape.
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/11 | 0/12 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/11 | 0/12 | 0/29

LIMITATIONS AND CAVEATS:
Limitations include a small sample size and the fact that we ceased recruitment to two of the treatment arms and changed our planned primary analysis mid-study based upon an interim analysis that was not specified at the time the study began.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No